CLINICAL TRIAL: NCT05083286
Title: A Randomized, Parallel-Group Study on the Duration Response of Highly Concentrated On Label Dose (COLD) of BOTOX® Compared to the On Label Dose and Concentration (OLD) in Subjects With Moderate to Severe Dynamic Glabellar Lines
Brief Title: Duration of Botox Using OLD Versus COLD for Treatment of Glabellar Lines
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Testing of Beverly Hills (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTBH-005
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Glabellar Frown Lines
Keywords: wrinkles; onabotulinumtoxinA
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- OLD (4 U per 0.1 mL) (Active Comparator): The total BOTOX dose will be 20U divided into 5 injections. Each injection will receive a total of 0.5 mL.
  Interventions: Drug: OnabotulinumtoxinA
- COLD (4 U per 0.02 mL group) (Active Comparator): The total BOTOX dose will be 20U divided into 5 injections. Each injection will receive a total of 0.1 mL.
  Interventions: Drug: OnabotulinumtoxinA

INTERVENTIONS:
Drug: OnabotulinumtoxinA — Injection of glabellar rhytids
  Other Names: Botox

SUMMARY:
This is a blinded, randomized study in the US to compare the duration response of two different concentrations of BOTOX in healthy female subjects with moderate to severe dynamic glabellar lines on maximum frown.

DETAILED DESCRIPTION:
This study involves a blinded, randomized, parallel-group design. The aim of this study is to evaluate the duration response of BOTOX in subjects with moderate to severe dynamic glabellar lines at the approved on-label dose of 20 U, however comparing the use of highly Concentrated On Label Dose (COLD) to the On Label Dose and concentration (OLD). The COLD concentration is defined as 4 Units per 0.02 mL and the OLD concentration is defined as 4 Units per 0.1 mL.

The total BOTOX dose will be 20U divided into 5 injections for both study groups. However, the injection volume will differ for the two study groups, such that the OLD (4 U per 0.1 mL) group will receive a total of 0.5 mL and the COLD (4 U per 0.02 mL) group will receive a total of 0.1mL.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of signing the informed consent.
* Overtly healthy as determined by medical evaluation (includes: medical history, physical examination, and vital signs).
* Subjects have moderate or severe dynamic glabellar lines on maximum frown as assessed with the Facial Wrinkle Scale.
* Female sex.
* Female subjects willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period. A female subject is eligible to participate if she is not pregnant (has a negative urine pregnancy result at Day 1 prior to treatment), is not breastfeeding, and at least one of the following conditions applies: 1) not a female of childbearing potential or 2) a female of childbearing potential who agrees to follow the contraceptive guidance.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form.
* Written informed consent from the subject has been obtained prior to any study-related procedures.
* Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable (eg, Written Authorization for Use and Release of Health and Research Study Information)
* Able, as assessed by the blinded evaluating investigator, and willing to follow study instructions and likely to complete all required study visits

Exclusion Criteria:

* Brow or eyelid ptosis, excessive dermatochalasis, deep dermal scarring, thick sebaceous skin, or an inability to substantially lessen upper facial rhytids, even by physically spreading them apart.
* Facial asymmetry including, in the opinion of the investigator, significant asymmetry with active contraction or at rest of the frontalis muscle.
* Medical condition that may increase the subject's risk of exposure to botulinum toxin, including diagnosed myasthenia gravis, Lambert-Eaton Syndrome, amyotrophic lateral sclerosis, or any other disease that might interfere with neuromuscular function.
* Profound atrophy/excessive weakness of muscles in target areas of injection.
* History of facial nerve palsy.
* Infection at the injection site or systemic infection.
* Presence of inflammation at the proposed injection site.
* Previous cosmetic surgery to the upper face (eg, periorbital surgery, brow lift, eyelid or eyebrow surgery), tissue grafting, or tissue augmentation with silicone or fat or other permanent fillers, or planning a facial cosmetic procedure during the study period.
* Subjects have been treated in the upper face (forehead lines, glabellar lines, crow's feet lines) within 1 year prior to the Baseline/Day 1 Visit with botulinum toxin therapy of any serotype.
* Noncompliance with the proper washout periods for prohibited medications/procedures.
* Subjects on topical retinoid therapy and/or topical hormone cream applied to the face, who have not been on a consistent dose regimen for at least 6 months prior to enrollment and who are unable to maintain a consistent dose regimen during the study.
* Oral retinoid therapy within 1 year prior to study enrollment.
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study.
* Females who are pregnant, breastfeeding, or planning a pregnancy during the study.
* Females of childbearing potential not using a reliable means of contraception.
* Known allergy or sensitivity to the study treatment or its components.
* Known immunization or hypersensitivity to any botulinum toxin serotype.
* Prior exposure to or anticipated need for treatment with botulinum toxin of any serotype for any reason during the study (other than study treatment).
* Evidence of recent alcohol or drug abuse.
* The subject has a condition or is in a situation which, in the investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Response Duration | 180 days
  Time to return to baseline Facial Wrinkle Scale (FWS) score at maximum frown, as assessed by the blinded evaluating investigator.
  The Facial Wrinkle Scale (FWS) scale ranges from a score of 0 to 3, and a higher score indicates greater (more severe) glabellar wrinkles.

SECONDARY OUTCOMES:
Investigator Live Assessment (Dynamic) | 180 days
  Responder rate at each visit on the Facial Wrinkle Scale (FWS) at maximum frown, as assessed by the blinded evaluating investigator.
  The responder rate is defined as the proportion of subjects maintaining a greater than or equal to 1 point improvement on the FWS.
  The Facial Wrinkle Scale (FWS) scale ranges from a score of 0 to 3, and a higher score indicates greater (more severe) glabellar wrinkles.
Subject Self Assessment (Dynamic) | 180 days
  Responder rate at each visit on the Facial Wrinkles Scale (FWS) at maximum frown, as assessed by the subject.
  The Facial Wrinkle Scale (FWS) scale ranges from a score of 0 to 3, and a higher score indicates greater (more severe) glabellar wrinkles.
Investigator Live Assessment (At Rest) | 180 days
  Responder rate at each visit on the Facial Wrinkle Scale (FWS) at rest, as assessed by the blinded evaluating investigator.
  The Facial Wrinkle Scale (FWS) scale ranges from a score of 0 to 3, and a higher score indicates greater (more severe) glabellar wrinkles.
Subject Self Assessment (At Rest) | 180 days
  Responder rate at each visit on the Facial Wrinkle Scale (FWS) at rest, as assessed by the subject.
  The Facial Wrinkle Scale (FWS) scale ranges from a score of 0 to 3, and a higher score indicates greater (more severe) glabellar wrinkles.
Change from Baseline Score | 180 days
  Change from baseline in mean Facial Wrinkle Scale (FWS) score at maximum frown, as assessed by the blinded evaluating investigator, at each visit.
  The Facial Wrinkle Scale (FWS) scale ranges from a score of 0 to 3, and a higher score indicates greater (more severe) glabellar wrinkles.
Change in Frontalis Function | 180 days
  Percentage of subjects with weakening of frontalis muscle function using the Frontalis Function Scale (FFS) compared to baseline, as assessed by the blinded evaluating investigator, at each visit.
  The Frontalis Function Scale (FFS) scale ranges from a score of 0 to 3, and a higher score indicates greater reduction of forehead movement during maximal brow raise.

CONTACTS AND LOCATIONS:
Overall Officials: John Joseph, MD, Principal Investigator — Clinical Testing of Beverly Hills
Locations (2):
- United States (2):
  - Clinical Testing of Beverly Hills, Encino, California
  - Steve Yoelin MD, Newport Beach, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blitzer A, Binder WJ, Aviv JE, Keen MS, Brin MF. The management of hyperfunctional facial lines with botulinum toxin. A collaborative study of 210 injection sites in 162 patients. Arch Otolaryngol Head Neck Surg. 1997 Apr;123(4):389-92. doi: 10.1001/archoto.123.4.389. PMID 9109785
- [Background] Carruthers A, Carruthers J, Said S. Dose-ranging study of botulinum toxin type A in the treatment of glabellar rhytids in females. Dermatol Surg. 2005 Apr;31(4):414-22; discussion 422. doi: 10.1111/j.1524-4725.2005.31107. PMID 15871316
- [Background] Carruthers JA, Lowe NJ, Menter MA, Gibson J, Nordquist M, Mordaunt J, Walker P, Eadie N; BOTOX Glabellar Lines I Study Group. A multicenter, double-blind, randomized, placebo-controlled study of the efficacy and safety of botulinum toxin type A in the treatment of glabellar lines. J Am Acad Dermatol. 2002 Jun;46(6):840-9. doi: 10.1067/mjd.2002.121356. PMID 12063480
- [Background] Carruthers J, Fagien S, Matarasso SL; Botox Consensus Group. Consensus recommendations on the use of botulinum toxin type a in facial aesthetics. Plast Reconstr Surg. 2004 Nov;114(6 Suppl):1S-22S. doi: 10.1097/01.PRS.0000144795.76040.D3. PMID 15507786